CLINICAL TRIAL: NCT03080766
Title: The Use of Decitabine as Induction Therapy for Acute Myeloid Leukemia With Complex and/or Monosomal Karyotype
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Principal Investigator, Dr. Anskar Y.H. Leung, Clinical Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML002
Record Dates: First submitted 2017-02-22; First posted 2017-03-15 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Acute Myeloid Leukemia; Complex Karyotype
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- decitabine (Experimental): Decitabine is a white to almost white powder for concentrate for solution for infusion. It is supplied as a lyophilized preparation in a clear colorless 20ml glass vial containing 50 mg decitabine.
  The concentrate should be aseptically reconstituted with 10 ml of water for injections. After reconstitution, the concentrate must be diluted within 15 minutes using cooled infusion fluids and completely administered to patients within 5 hours.
  The drug will then be administrated intravenously.
  Dosage 20 mg/m2
  28-day course, for each course, receive decitabine for 10 days
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — Decitabine (trade name Dacogen®) is a cytidine deoxynucleoside analogue, which selectively inhibits DNA methyltransferases at low doses, resulting in gene promoter hypomethylation that can result in reactivation of tumor suppressor genes, induction of cellular differentiation or cellular senescence followed by programmed cell death.
  Other Names: Dacogen

SUMMARY:
Acute myeloid leukemia (AML) is a heterogeneous group of diseases with distinct clinicopathologic features sharing in common an abnormal increase in myeloblasts in blood and bone marrow (BM). In about 5-10% patients, the myeloblasts exhibit chromosomal abnormalities (complex and/or monosomal karyotype, CK/MK*) that are associated with refractoriness to conventional chemotherapy and an extremely bad prognosis.

Standard induction chemotherapy for AML comprises daunorubicin and cytarabine, the "7+3" regimen. However, treatment is largely ineffective for CK/MK AML with a temporary clearance of blasts achieved in only 30-40% cases and the cumulative toxicities resulting from repeated courses of chemotherapy have significantly increased the morbidity and mortality risks in subsequent allogeneic BMT. Therefore, standard treatment is unsatisfactory and there is an unmet clinical need for more effective and less toxic induction regimen.

Both previous and recent studies showed that 10 day course of decitabine (20 mg/m2/day) induced remission in 70-100% patients with CK/MK AML, particularly those with TP53 mutations. In this study, patients with CK/MK AML will be treated with decitabine to induce remission. Bone marrow examination will be performed after each course until complete clearance of blasts or disease progression. Patients achieving CR/CRi (see below) will continue to receive 4 more courses, after which patients eligible for BMT and for whom donors are available will receive curative BMT. We reckon that the time it takes for 4 courses of decitabine will suffice for transplantation workup in HK. . Patients ineligible for BMT will continue to receive decitabine until leukemia progression. The response rate, leukemia free survival (LFS), overall survival (OS) and percentage of patients who can be bridged to BMT will be compared with historical 7+3 regimen control.

DETAILED DESCRIPTION:
This is an open-label interventional study to study the use of decitabine as induction therapy for acute myeloid leukemia with complex and/or monosomal karyotype.

Subjects will receive decitabine for every 28 days, until disease progression or a bone marrow transplantation is carried out, in the schedule as below:

Cycle 1:

Receive decitabine for 10 days

Cycle 2 and Cycle 3:

Based on the result of bone marrow examination, subjects may receive decitabine for 5 days or 10 days

Cycle 4 until disease progression:

Rdecitabine for 5 days. Subjects may also resume a 10 day treatment after cycle 6 if their physician judged as appropriate.

The drug will then be administrated intravenously.

Blood will be drawn every 7 days and bone marrow extraction would be done on Day 28 (+/- 3days) from the day 1 of each cycle of treatment for examination.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age 18-65 years old) with CK/MK AML at diagnosis
2. De novo or secondary AML is allowed
3. ECOG performance ≤ 2
4. Subjects with adequate liver, pancreatic and renal function at screening as demonstrated by :Direct bilirubin < 2 x upper limit of laboratory normal (ULN) Alanine aminotransferase (ALT) < 2.5 x ULN MDRD-eGRF > 30ml/min/1.73m2
5. Negative serum / urine pregnancy test within 7 days before starting study treatment in women with childbearing potential.
6. Subjects with ability to understand the protocol and signed a written informed consent document prior to the participation of the study.

Exclusion Criteria:

1. Patients with CK/MK AML who have received standard induction chemotherapy before
2. Patients with active and uncontrolled infection.
3. Patients with concurrent severe and uncontrolled concomitant medical conditions that could cause unacceptable safety risk or compromise compliance with the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-28 (Estimated)

PRIMARY OUTCOMES:
Complete remission (CR): | up to 16 weeks
  No increase in blasts in BM or PB (<5% of total nucleated cells), with absolute neutrophil count ≥ 1x109/L and platelet count ≥ 100 x109/L.

CONTACTS AND LOCATIONS:
Overall Officials: Anskar Leung, Professor, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided